CLINICAL TRIAL: NCT00956371
Title: A Double-Blind, Placebo-Controlled, SIngle Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-7746 in Healthy Adult Subjects
Brief Title: ONO-7746 Study in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-7746POU001
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-7746; Healthy adult subjects

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- P (Placebo Comparator)
  Interventions: Drug: ONO-7746
- E (Experimental)
  Interventions: Drug: ONO-7746

INTERVENTIONS:
Drug: ONO-7746 — 5mg, 10mg, 20mg, 50mg, 100mg, 200mg, 400mg, 800mg, 1200mg QD/1 day
  Arms: P
Drug: ONO-7746 — 5mg, 10mg, 20mg, 50mg, 100mg, 200mg, 400mg, 800mg, 1200mg QD/1 day
  Arms: E

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ONO-7746 in healthy adult subjects. The secondary objectives are to characterize the pharmacokinetic and pharmacodynamic profiles of ONO-7746.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male or female subjects (18-55 years inclusive)
* Body mass index (BMI) of 19-35 kg/m² (inclusive)
* For females: postmenopausal, non-lactating and non-pregnant

Exclusion Criteria:

* History or presence of clinically significant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-7746 across ascending single doses | study duration

SECONDARY OUTCOMES:
Characterization of PK and PD profiles of ONO-7746 | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Austin, Austin, Texas, United States